CLINICAL TRIAL: NCT05642728
Title: Impact of a Personalised Tele-case Management Follow-up Programme on Asthma Control, Exacerbations and Use of Healthcare Resources in Moderate and Severe Asthmatics: PERCASTHMA Study.
Brief Title: Impact of a PERsonalized CAse MAnagement Program for the Follow-up of Moderate and Severe aSTHma Patients on Exacerbations, Health Resource Use and Asthma Control: PERCASTHMA STUDY
Acronym: PERCASTHMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MurciaSalud (Other Government)
Responsible Party: Principal Investigator, Manuel Castilla Martinez, Principal Investigator, MurciaSalud
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PERCASTHMA STUDY
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Asthma; Case Management; Telemedicine
Keywords: asthma; case manager; telemedicine; exacerbations
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case management group (Experimental)
  Interventions: Other: Case management follow-up program
- Control group (No Intervention)

INTERVENTIONS:
Other: Case management follow-up program — The case manager will monitor asthma control (asthma control test, ACT) and adherence to treatment with questionnaires (inhaler adherence test, TAI) and electronic prescription withdrawal (e-prescription). The case manager will make decisions based on these results and according to pre-designed medical instructions. In addition, the patient will be able to contact the case manager for advice during periods of worsening symptoms. The patient will contact the case manager via a mobile app with messaging and video call option, as well as a contact phone number and email for consultations.
  Arms: Case management group

SUMMARY:
The goal of this randomized clinical trial is to learn about the impact of the implementation of an intervention-based case management follow-up program during periods of clinical worsening or poor adherence in patients with moderate and severe asthma.

Patients will be randomized into two arms: a case management follow-up group and a control group that will follow-up according to routine care practice. A single masking (outcomes assessor) was performed. Researchers will compare the response on exacerbations, health resource use and asthma control between the two groups during a one-year follow-up. Outcomes on pulmonary function, quality of life, adherence to treatment, pulmonary inflammation parameters and systemic corticosteroid use will also be studied. Additionally, other baseline clinical characteristics and events of the previous year will be collected retrospectively for all patients.

The study was evaluated and approved by a local ethics committee.

All study participants will receive an asthma education session with review of inhaler technique and training in the use of self-management action plans. Only participants in the case management follow-up group will periodically send asthma control (ACT) and adherence (TAI) questionnaires to the case manager. If not completed, the case manager will contact the patient by telephone to determine the degree of asthma control and adherence. The case manager will also monitor the withdrawal of drugs on the electronic prescription. The patient will contact the case manager via a mobile app, phone or email if needed due to worsening symptoms or need for self-management support. With this information, the case manager will make decisions based on personalized medical instructions prepared by the pulmonologist at the baseline visit, which will be reviewed according to evolution.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Previous diagnosis of bronchial asthma according to GEMA 5.4 criteria.

  • Follow-up for at least 6 months in an asthma unit and absence of relevant uncontrolled comorbidities.
* Classified as moderate or severe asthma according to therapeutic step at the beginning of the study, as defined by GEMA 5.4.
* Signed informed consent form.

Exclusion Criteria:

* Simultaneous presence of other diseases that may simulate asthma symptoms (COPD, left heart failure, functional dyspnea/hyperventilation syndrome, inducible laryngeal obstruction...).
* Severe psychosocial problems or any other clinical situation that prevents the signature of the informed consent and/or the follow-up proposed in the study.
* Lack of minimum technological knowledge for the use of monitoring tools.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Median ACT score at 6 and 12 months compared with control group and baseline | At 6 and 12 months
  ACT is a validated, self-administered questionnaire to assess asthma control in the last 4 weeks. Possible scores range from 5 (worst possible control) to 25 (best possible control). Scores equal to or greater than 20 suggest good asthma control. Median ACT score at 6 and 12 months compared with control group and baseline
Median of total and severe exacerbations at 12 months | From baseline to 12 months
  Hospital admissions, emergency room visits, and unscheduled medical visits for asthma exacerbation accumulated at the end of the follow-up period compared with control group and baseline
Median healthcare resources use at 12 months | From baseline to 12 months
  Healthcare resource use was defined as the addition of the number of unscheduled medical visits in primary care, emergency department care and hospitalisations. Median use of health resources at 12 months compared with control group and baseline

SECONDARY OUTCOMES:
Median of electronic prescription withdrawal at 12 months | At 12 months
  To assess adherence, the percentage of withdrawal of inhaled glucocorticoid e-prescriptions will be measured.
Median pre-bronchodilator forced expiratory volume in the first second (pre-bronchodilator FEV1) and zscore at 6 and 12 months | At 6 and 12 months
  Lung function was measured according to the SEPAR guidelines. Zscore is a tool to express results of spirometry that facilitates interpretation and comparison between patients with different characteristics. The Z-score indicates how many standard deviations a measured value is from predicted. Median pre-bronchodilator forced expiratory volume in the first second (pre-bronchodilator FEV1) and zscore at 6 and 12 months compared with control group and baseline
Median AQLQ score at 6 and 12 months | At 6 and 12 months
  Asthma Quality of Life Questionnaire (AQLQ) is a validated, self-administered questionnaire to assess quality of life related to asthma. Possible scores range from 1 (worst possible quality of life) to 7 (best possible). The minimum clinically significant change is 0.5 points. Median AQLQ score at 6 and 12 months compared with control group and baseline.
Median FeNO value at 6 and 12 months | At 6 and 12 months
  Exhaled nitric oxide (FeNO) will be measured using NioxVero electrochemical analyser according to standard use technique. FeNO is measured in ppb. Median FeNO value at 6 and 12 months compared with control group and baseline.
Median blood eosinophil count at 12 months | At 12 months
  Median blood eosinophil count at 12 months compared with control group and baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Los Arcos del Mar Menor, San Javier, Murcia, Spain